CLINICAL TRIAL: NCT04917146
Title: "Family Caregiver Reflex": Family Support for Patients Followed for Systemic Sclerosis - Pilot Study Evaluating the Experience and Role of Family Caregivers in Order to Identify and Include Them in Therapeutic Educational Programs
Brief Title: Systemic Sclerosis' Relatives Reflex
Acronym: RelativReflex
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: FSMR FAI2R (Unknown); Ministère des solidarités et de la santé (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210756
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Systemic Sclerosis; Caregivers
Keywords: Systemic sclerosis; Relatives caregivers; Therapeutic education program
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers (CG): Caregivers of patients with systemic Scleroderma
  Interventions: Other: Self-administered questionnaires for relatives (caregivers=CG)

INTERVENTIONS:
Other: Self-administered questionnaires for relatives (caregivers=CG) — Sociodemographic and medical information for the patient and the CG. SF36 questionnaire for the quality of life (physical, mental) of family CGs This assessment will be supplemented by specific questions relating to: physical health, emotional state, personal and leisure activities of the caregiver.
  The CG's knowledge and representations of the disease : questions adapted from the Brief-IPQ disease representation questionnaire.
  Questions will also focus on the caregiver's reactions to the patient's illness.
  We have constructed a questionnaire to assess the main areas of aid in the context of SSc: emotional, domestic help, administrative, medical, for trave (16 items and an open question).
  The CG Reaction Assessment-CRA questionnaire to assess the positive and negative dimensions of helping (24 items). It assesses five dimensions: self-esteem, financial impact, impact on health, impact on time and lack of family support.
  The reason for the assistance provided.

SUMMARY:
Systemic sclerosis (SSc) is a rare, serious disease that is part of chronic inflammatory rheumatism.

It requires multidisciplinary care and a specific therapeutic patient education program.

SSc actually affects every member of the family, the patient as well as those close to him. It deeply affects each member of the family (increased fatigue, stress, social isolation, exhaustion, financial difficulties …) which gives rise to threats of vulnerability and modulates the balance of family relations.

However, there are very few studies on family SSc caregivers. We have raised the question about the experience and needs of caregivers in order to better support them.

The main purpose of this pilot study is to better understand the particularities of relatives (caregivers) of patients suffering from systemic sclerosis and will allow us to refine our knowledge about the assistance they provide for SSc patients and its impact on family caregivers :

* lived experience of the relatives (caregivers);
* physical, mental and socio-professional health of the relatives (caregiver);
* relationship between the relative (caregiver) and the patient.

The research will be carried out at Cochin Hospital, in collaboration with the French Scleroderma Association (ASF).

It will be offered to relatives of SSc patients identified by health team in the rheumatology or internal medicine department, as well as during consultations and patient education activities.

An information note and an informed consent will be given to each patient and his caregiver ; Self-questionnaires will then be offered to relatives.

They can fill them out while they are in the hospital, or at home and return the completed questionnaire.

Caregivers will be questioned about their quality of life, health, relationship with the patient and support situation.

They will also be asked for personal socio-demographic information concerning the patient.

The "caregiver reflex" project is part of the 2020-2022 mobilization and support strategy for caregivers "acting for the health of family caregivers", in which the establishment of a "caregiver reflex" among professionals health is put forward.

DETAILED DESCRIPTION:
Exploratory study with family caregivers of patients suffering from Systemic Sclerosis (SSc).

This research work will allow to better understand the experiences and needs of these very particular caregivers, in order to offer them specific educational support and workshops.

It should also allow healthcare teams to develop a "family caregiver reflex", especially in the context of SSc disease to identify and include PAs in PTE programs.

Primary objectives:

Identify caregivers in the SCS patient's family circle: in order to analyze their profile and assess their needs, expectations, projects and difficulties:

* Identify who are the caregivers of SSc people: epidemiological data, profiles of SSc patients followed in rheumatology and Internal medicine departments of Cochin hospital (sex, age, professional activity, possible presence of young people in the entourage, etc.);
* assess the assistance provided by the caregivers: type and specificity;
* Specify the experience and feelings of the caregivers in relation to this aid (positive or negative impact)
* Identify fragile-vulnerable caregivers .

Secondary objectives:

Develop, from this data, educational tools to share with the other members of the FSMR FAI2R and specifically dedicated to the caregivers of SSc patients:

* "Caregiver reflex" tool intended for professionals to better identify and identify caregivers of SSc patients;
* Specific interview guide for the educational diagnosis of caregivers;
* Examples of educational workshops for caregivers meeting identified needs (workshop experienced by the illness of the other, stress management, fatigue, dietary advice, lifestyle, to assist persons in administrative and social procedures...)

ELIGIBILITY:
Inclusion Criteria:

* Relatives caregivers of patients suffering from Systemic Scleroderma (family, friends, neighbours);
* Be at least 18 years old;
* Not being the patient's professional caregiver;
* Have signed the informed consent to participate.

Exclusion Criteria:

* Inability to answer questionnaires (language, cognitive disorders, etc.).
* under curatorship or tutorship
* with State medical care (AME)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants:
  relatives of patients suffering from Systemic Scleroderma
  Two possible inclusion methods:
  1. At the hospital, via health professionals (doctor, nurse, social worker, etc.) who identify the loved one accompanying the patient during a consultation or hospitalization;
  2. Via the French Scleroderma Association - ASF (call for participation)
  They will be presented with the study by the recruiting psychologist or education nurse and given an information note and consent to participate. Patients will also be presented with an information letter and consent to participate .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Inclusion visit 1 day
  Sociodemographic and medical information concerning the patient assisted Patients' sociodemographic and medical information will be collected: age, gender, family composition, family relationship with the family caregiver, length of the illness.

SECONDARY OUTCOMES:
Questionnaire | Inclusion visit 1 day
  Socio-demographic information about the caregiver Sociodemographic information will be collected on the informal caregiver: age, sex, professional situation, seniority of the help.
Questionnaire SF36 | Inclusion visit 1 day
  Physical and mental health The SF36 questionnaire (Leplège et al., 1998) will be used to assess the quality of life of family caregivers.
  This widely used questionnaire is divided on 6 items assessing the physical and mental quality of life.
  This assessment will be supplemented by specific questions relating to:
  * Physical health: presence of chronic pathologies, medical monitoring, taking treatment, health behaviors (diet, tobacco, alcohol);
  * The emotional state;
  * The personal and leisure activities of the caregiver.
Questionnaire | Inclusion visit 1 day
  The relationship with the patient The caregiver's knowledge and representations of the disease will be assessed using questions adapted from the Brief-IPQ disease representation questionnaire (Broadbent et al., 2006).
  Questions will also focus on the caregiver's reactions to the patient's illness.
Questionnaire | Inclusion visit 1 day
  Aid activities To date, there is no questionnaire to assess the aid activity in the context of chronic inflammatory rheumatism. The existing questionnaires on the subject being too often linked to situations of significant dependence, as in the context of neurodegenerative diseases, we have constructed a questionnaire to assess the main areas of aid in the context of SSc: emotional, domestic help , administrative, medical, for travel. It is composed of 16 items and an open question.
Questionnaire | Inclusion visit 1 day
  Positive and negative dimensions of aid The Caregiver Reaction Assessment-CRA questionnaire (Given et al., 1992) will be used to assess the positive and negative dimensions of helping. This questionnaire has 24 items. It assesses five dimensions: self-esteem, financial impact, impact on health, impact on time and lack of family support.
  Finally, two questions are asked to assess the reason for the assistance provided.

CONTACTS AND LOCATIONS:
Overall Officials: Janine-Sophie Giraudet-Le Quintrec, MD, Principal Investigator — Cochin Hospital - APHP
Locations (1):
- Rhumatology Service, Paris, France

REFERENCES:
- [Background] Brignon M, Vioulac C, Boujut E, Delannoy C, Beauvais C, Kivits J, Poivret D, Giraudet Le Quintrec JS, Untas A, Rat AC. Patients and relatives coping with inflammatory arthritis: Care teamwork. Health Expect. 2020 Feb;23(1):137-147. doi: 10.1111/hex.12982. Epub 2019 Nov 27. PMID 31774612
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Brouwer WB, van Exel NJ, van de Berg B, Dinant HJ, Koopmanschap MA, van den Bos GA. Burden of caregiving: evidence of objective burden, subjective burden, and quality of life impacts on informal caregivers of patients with rheumatoid arthritis. Arthritis Rheum. 2004 Aug 15;51(4):570-7. doi: 10.1002/art.20528. PMID 15334429
- [Background] Canedo-Ayala M, Rice DB, Levis B, Carrier ME, Cumin J, Malcarne VL, Hagedoorn M, Thombs BD; Scleroderma Caregiver Advisory Committee. Factors associated with symptoms of depression among informal caregivers of people with systemic sclerosis: a cross-sectional study. Disabil Rehabil. 2020 Feb;42(3):394-399. doi: 10.1080/09638288.2018.1500647. Epub 2018 Aug 19. PMID 30122129
- [Background] Given CW, Given B, Stommel M, Collins C, King S, Franklin S. The caregiver reaction assessment (CRA) for caregivers to persons with chronic physical and mental impairments. Res Nurs Health. 1992 Aug;15(4):271-83. doi: 10.1002/nur.4770150406. PMID 1386680
- [Background] Jacobi CE, van den Berg B, Boshuizen HC, Rupp I, Dinant HJ, van den Bos GA. Dimension-specific burden of caregiving among partners of rheumatoid arthritis patients. Rheumatology (Oxford). 2003 Oct;42(10):1226-33. doi: 10.1093/rheumatology/keg366. Epub 2003 Jun 16. PMID 12810934
- [Background] Kasle S, Wilhelm MS, Zautra AJ. Rheumatoid arthritis patients' perceptions of mutuality in conversations with spouses/partners and their links with psychological and physical health. Arthritis Rheum. 2008 Jul 15;59(7):921-8. doi: 10.1002/art.23821. PMID 18576302
- [Background] Lam M, Lehman AJ, Puterman E, DeLongis A. Spouse depression and disease course among persons with rheumatoid arthritis. Arthritis Rheum. 2009 Aug 15;61(8):1011-7. doi: 10.1002/art.24510. PMID 19644902
- [Background] Leplege A, Ecosse E, Verdier A, Perneger TV. The French SF-36 Health Survey: translation, cultural adaptation and preliminary psychometric evaluation. J Clin Epidemiol. 1998 Nov;51(11):1013-23. doi: 10.1016/s0895-4356(98)00093-6. PMID 9817119
- [Background] Matheson L, Harcourt D, Hewlett S. 'Your whole life, your whole world, it changes': partners' experiences of living with rheumatoid arthritis. Musculoskeletal Care. 2010 Mar;8(1):46-54. doi: 10.1002/msc.165. PMID 20077577
- [Background] Rice DB, Canedo-Ayala M, Carboni-Jimenez A, Carrier ME, Cumin J, Malcarne VL, Hagedoorn M, Thombs BD; Scleroderma Caregiver Advisory Team. Challenges and support service preferences of informal caregivers of people with systemic sclerosis: a cross-sectional survey. Disabil Rehabil. 2020 Aug;42(16):2304-2310. doi: 10.1080/09638288.2018.1557268. Epub 2019 Jan 29. PMID 30696293
- [Background] Untas A, Vioulac C, Boujut E, Delannoy C, Poivret D, Rat AC, Beauvais C, Giraudet Le Quintrec JS. What Is Relatives' Role in Arthritis Management? A Qualitative Study of the Perceptions of Patient-Relative Dyads. Patient Prefer Adherence. 2020 Jan 7;14:45-53. doi: 10.2147/PPA.S231919. eCollection 2020. PMID 32021116